CLINICAL TRIAL: NCT04176380
Title: Phase II Trial of Autologous Rapamycin-Resistant Th1/Tc1 (RAPA-201) Cell Therapy of Relapsed, Refractory Multiple Myeloma
Brief Title: RAPA-201 T Cell Therapy for Relapsed, Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rapa Therapeutics LLC (Industry)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPA-201-RRMM
Record Dates: First submitted 2019-11-12; First posted 2019-11-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Relapsed, Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Autologous Th1/Tc1 cell Therapy; RAPA-201
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of RAPA-201 cells (Experimental)
  Interventions: Biological: RAPA-201 Autologous T cells

INTERVENTIONS:
Biological: RAPA-201 Autologous T cells — Autologous rapamycin resistant Th1/Tc1 cells
  Other Names: RAPA-201 cells

SUMMARY:
RAPA-201-RRMM is an open-label, single-arm, non-randomized multicenter phase II study of RAPA-201 autologous T cells in adults with relapsed, refractory multiple myeloma who have received at least three (3) prior lines.

DETAILED DESCRIPTION:
This clinical trial evaluates autologous rapamycin-resistant Th1/Tc1 (RAPA-201) cells for therapy of relapsed, refractory multiple myeloma (RRMM). The study population of RRMM patients is defined by: relapse after ≥ 3 prior regimens; exposure to ≥ 2 proteasome inhibitors (PI) (e.g. bortezomib), ≥ 2 immunomodulatory agents (IMiD) (e.g. lenalidomide), and ≥ 1 anti-CD38 monoclonal antibody (e.g., daratumumab); and refractory status to ≥ 1 PI agent and ≥ 1 IMiD agent. The primary study objective is to determine the overall response rate, as evaluated by IMWG criteria, of RAPA-201 cells and a pentostatin-cyclophosphamide (PC) host conditioning regimen in patients with RRMM. A sample size of 22 patients was selected to determine whether RAPA-201 therapy represents an active regimen in RRMM, as defined by a response rate (≥ partial remission) consistent with a 35% rate.

Multiple myeloma (MM) is an incurable cancer characterized by clonal proliferation of plasma cells. MM is the second most common form of hematologic malignancy in the United States, with approximately 11,000 individuals dying from the disease in 2014. Due in part to the aging population, MM prevalence will dramatically increase in the next few decades. MM management has many FDA-approved options for the up-front setting, maintenance therapy, and therapy at second or third relapse. For patients with relapsed MM, therapy typically consists of triplet regimens approved by the U.S. Food and Drug Administration (FDA), including the KRd, DRd, and DPd regimens. Although triplet regimens are improved relative to prior therapies, they typically provide a progression-free survival of less than two years and cause substantial toxicities. Few standard, effective options exist for patients with MM who have more advanced disease and higher levels of drug refractoriness. In contrast to drug and monoclonal antibody therapy, which are essentially non-curative, T cell therapy can cure MM, as evidenced by long- term survival in recipients of allogeneic hematopoietic cell transplantation. The promise of T cell therapy against MM is further exemplified by high response rates using gene-modified autologous CAR-T cell therapy directed against the BCMA target. However, CAR-T therapy is limited by variable tumor cell target expression, which compromises response durability leading to relapse. Furthermore, CAR-T cell products are expensive to manufacture, with the financial burden further complicated by frequent inpatient hospital monitoring and treatment of potentially lethal toxicities that include cytokine storm and neurologic damage. Thus, a great need exists to develop novel T cell therapies for RRMM that are safe, cost effective, and curative. We will evaluate one such promising candidate, namely, autologous rapamycin-resistant Th1/Tc1 cells (RAPA-201).

RAPA-201 cell therapy differs from existing approaches in several important categories. First, RAPA-201 cells are rendered rapamycin-resistant by proprietary ex vivo manufacturing that rapidly and cost effectively de- differentiates senescent patient T cells, which results in a therapeutic product enriched for the beneficial T central memory (TCM) subset and severely depleted of checkpoint inhibitory receptors that inhibit anti-cancer effects. This depth and breadth of T cell re-programming is not possible in vivo due to toxicity of pharmacologic agents, which can be rendered completely non-toxic through drug extracorporealization. Operating together, T cell rapamycin-resistance, TCM differentiation, and checkpoint removal promotes RAPA-201 T cell in vivo persistence and in vivo activity required for curative anti-tumor effects. Second, RAPA-201 cells are manufactured in a high, otherwise toxic dose of the critical anti-cancer cytokine IFN-α, which promotes a CD4+Th1 and CD8+Tc1 T cell phenotype that optimizes anti-tumor effects. Third, rapamycin-resistant T cells express a diverse T cell receptor repertoire that can address the complex biology of multiple myeloma, where tumor antigens are either not known or variable over time due to tumor genetic instability. Because polyclonal RAPA-201 T cells are capable of in vivo expansion to tumor antigens, RAPA-201 therapy can be applied not only to RRMM but also to other hematologic malignancies and common solid tumors, including lung cancer resistant to PD(L)-1 checkpoint therapy. And fourth, RAPA-201 cell therapy will be administered in combination with a novel host conditioning regimen consisting of pentostatin and low-dose, dose-adjusted cyclophosphamide (PC regimen). The PC regimen causes host lymphoid depletion while sparing host myeloid cells, thus permitting repeat therapeutic RAPA-201 cycles in the outpatient setting with reduced financial burden and without substantial neutropenia and associated opportunistic infection. As such, the PC regimen safely creates "immune space" in the RRMM patient, thereby potentiating the in vivo expansion and curative potential of RAPA-201 cells.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Diagnosis of relapsed, refractory multiple myeloma.
* Exposure to at least three different prior lines of therapy including exposure to at least two proteosome inhibitors (e.g. bortezomib), and at least two immunomodulatory drugs (e.g. lenalidomide) and at least one anti-CD38 monoclonal antibody agent (e.g. daratumumab). To qualify as a prior line of therapy, ≥ 2 cycles of therapy must be administered unless the disease is refractory, or the regimen is not tolerated. Documentation of a prior line of therapy must include at least one of the following three items: [1] medical records detailing prior treatment, best response to treatment, and date of progression; [2] myeloma markers (SPEP, UPEP, Immunoglobulin, FLC) at time of treatment and progression; or, [3] documentation by investigator/treating physician to be included in patient's medical and research record (for example, note in electronic medical record), indicating prior treatment, best response to treatment, and data of progression.
* Refractory status to ≥ one proteasome inhibitor AND ≥ one immunomodulatory drug. Refractory disease is defined as <25% reduction in M-protein/free light chain difference (involved vs. uninvolved) or disease progression during treatment or ≤ 60 days after treatment cessation. Patient may or may not be refractory to anti-CD38 therapy.
* Presence of secretory myeloma/measurable disease, as defined by ONE of the following:

  1. Serum M-protein (SPEP) ≥ 0.5 mg/dL or
  2. Urine M-protein (UPEP) ≥ 200 mg/24 hours; or
  3. Light chain MM: Serum free light chain (FLC) assay ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa/lambda FLC ratio.
* Must have a potential source of autologous T cells potentially sufficient to manufacture RAPA-201 cells, as defined by a circulating CD3+ T cell count ≥ 300 cells/µL.
* Prior to apheresis, patients must be ≥ 14 calendar days from last myeloma therapy, major surgery, radiation therapy and participation in investigational trials.
* Patients must have recovered from clinical toxicities (resolution of CTCAE toxicity to a value of ≤ 2).
* Left ventricular ejection fraction (LVEF) by MUGA or 2-D echocardiogram within institution normal limits, with an LVEF level of ≥ 40%.
* Serum creatinine ≤ to 2.5 mg/dL.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ to 3 x upper limit of normal (ULN).
* Absolute neutrophil count (ANC) of ≥ 1000 cells/µL (independent of growth factor support for at least 7 days prior to screening).
* Platelet count of ≥ 50,000 cells/µL, with value obtained (independent of growth factor support or transfusion support for at least 7 days prior to screening).
* Hemoglobin count ≥ 8 grams/µL (independent of growth factor support or transfusion support for at least 7 days prior to screening).
* Bilirubin ≤ 1.5 (except if due to Gilbert's disease).
* Corrected DLCO ≥ 50% (Pulmonary Function Test).
* No history of abnormal bleeding tendency, as defined by any inherited coagulation defect or history of internal bleeding.
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior allogeneic stem cell transplantation.
* Current plasma cell leukemia (circulating myeloma > 20% of leukocytes).
* Other active malignancy (except for non-melanoma skin cancer).
* Non-secretory multiple myeloma (difficult to assess by IMWG criteria).
* Evidence of systemic AL Amyloidosis involving any vital organ. Incidental histologic demonstration of amyloid deposition in marrow/within plasmacytoma is not considered organ involvement.
* Life expectancy <4 months.
* Patients seropositive for HIV, hepatitis B, or hepatitis C.
* Uncontrolled hypertension.
* History of cerebrovascular accident within 6 months prior to enrollment.
* Myocardial infarction within 6 months prior to enrollment.
* NYHA class III/IV congestive heart failure.
* Uncontrolled angina/ischemic heart disease.
* Subjects with known central nervous system disease.
* Pregnant or breastfeeding patients.
* Patients of childbearing age, or males who have a partner of childbearing potential, who are unwilling to practice contraception.
* Patients may be excluded at PI discretion or if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | One (1) year after last dose of RAPA-201 cells.
  To determine the overall response rate, as evaluated by IMWG criteria, in patients with relapse, refractory multiple myeloma (RRMM) treated with autologous RAPA-201 cells and a pentostatin-cyclophosphamide (PC) host conditioning regimen.

SECONDARY OUTCOMES:
Effect of therapy on disease control | One (1) year after the last dose of RAPA-201 cells.
  (1) To determine the effect of therapy on multiple myeloma disease control, including duration of response (DOR; time from initial tumor response to disease progression).
Effect in Quality of Life | One (1) year after the last dose of RAPA-201 cells.
  To evaluate the effect of therapy on quality of life (QOL) using the FACT-BMT survey.

OTHER OUTCOMES:
Immune reconstitution | Screening; Day 1 of every treatment cycle; End of treatment; Day 1 of Months 1, 3, 9 and 12 of Follow-up.
  Immune reconstitution of participants receiving RAPA-201 cells will be measured using flow cytometry to obtain the absolute number of circulating CD4+ and CD8+ T cells per microliter of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fowler, M.D., Study Director — Rapa Therapeutics LLC
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhakal B, Hari P, Chhabra S, Szabo A, Lum LG, Glass DD, Park JH, Donato M, Siegel DS, Felizardo TC, Fowler DH. Rapamycin-resistant polyclonal Th1/Tc1 cell therapy (RAPA-201) safely induces disease remissions in relapsed, refractory multiple myeloma. J Immunother Cancer. 2025 Jan 28;13(1):e010649. doi: 10.1136/jitc-2024-010649. PMID 39875173